CLINICAL TRIAL: NCT06531733
Title: Sleep and Wake Countermeasures for Artemis: In-laboratory Study
Brief Title: Artemis Sleep Countermeasures
Acronym: ASCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erin E. Flynn-Evans, Fatigue Countermeasures Laboratory Director, National Aeronautics and Space Administration (NASA)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000748
Record Dates: First submitted 2024-06-07; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: 8 participants per condition (24 total across 3 conditions + 1 sham/placebo condition that everyone will experience)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sleep promoting + wake placebo (Experimental): Participants in this condition will listen to pink noise during a sleep opportunity (sleep promoting) and then have normal light with no nap (sham/placebo).
  Interventions: Device: Sleep Promoting (pink noise); Device: Wake Promoting (blue enriched light plus a nap)
- sleep placebo + wake promoting (Experimental): Participants in this condition will have a sleep opportunity with no pink noise (sham/placebo) and then be exposed to blue enriched light (wake promoting) after a nap.
  Interventions: Device: Sleep Promoting (pink noise); Device: Wake Promoting (blue enriched light plus a nap)
- sleep promoting + wake promoting (Experimental): Participants in this condition will be exposed to pink noise during a sleep opportunity (sleep promoting) and then be exposed to blue enriched light (wake promoting) after a nap.
  Interventions: Device: Sleep Promoting (pink noise); Device: Wake Promoting (blue enriched light plus a nap)

INTERVENTIONS:
Device: Sleep Promoting (pink noise) — Participants will be provided with comfortable headphones to wear throughout their daytime sleep opportunity. The headphones will deliver a continuous pink noise sound no greater than 50 decibels. Participants will be allowed to turn down the sound of the pink noise if they find it too loud. Participants will wear the headphones with no noise during the placebo condition.
Device: Wake Promoting (blue enriched light plus a nap) — Participants randomized to the blue-enriched light and nap condition will have the blue-enriched light turned on during their nighttime stay in the lab. The light will be turned off for up to one hour during the nap. During the placebo condition, participants will have an overhead room light of ~150 lux illuminated throughout their nighttime stay in the lab. This light level reflects an older NASA standard which was used in the design of some Artemis vehicles. During the placebo condition, participants will be asked to engage in quiet activities such as reading for one hour.

SUMMARY:
Purpose. The purpose of this study is to test sleep and wake-promoting countermeasures to evaluate their effectiveness in helping individuals fall asleep quickly, maintain sleep during a nap, and maintain alertness during waking.

Protocol Overview. The proposed study involves two laboratory visits separated by at least one week. Participants are required to complete all procedures in the companion screening and at-home protocol in order to qualify for this laboratory protocol. The at-home protocol involves keeping a regular schedule for 2-3 weeks. Participants will need to maintain a regular schedule with at least 8.5 hours in bed for at least one week prior to the first laboratory visit. They will then continue the at-home protocol, maintaining at least 8.5 hours in bed each night for at least a week before completing the second laboratory visit.

There are two interventions that participants will experience during the study, sleep promoting (pink noise) and wake promoting (blue enriched lighting plus a nap). These will be delivered separately and together depending on randomization.

Participants will first be randomized to one of three conditions sleep promoting + wake placebo, sleep placebo + wake promoting, or sleep promoting + wake promoting. All participants will complete a sleep placebo + wake placebo condition. The order of the full placebo condition versus the intervention (i.e., lab visit 1 vs. lab visit 2) will be randomized after the condition randomization occurs. Each participant will complete one of the interventions and one placebo for a total of two visits.

DETAILED DESCRIPTION:
SPECIFIC AIMS The investigators aim to test whether pink noise can improve sleep outcomes and subsequent alertness. The investigators further aim to test whether pink noise induced sleep improves alertness and performance during the night alone or in combination with blue-enriched lighting and a nap. Finally, the investigators will test whether blue-enriched lighting and a nap can improve alertness and performance during the night.

HYPOTHESES

1. The investigators hypothesize that exposure to pink noise during a daytime sleep opportunity will improve sleep onset latency, sleep duration, and sleep depth compared to a control condition with no noise.
2. The investigators hypothesize that sleep induced by pink noise will improve subjective alertness and performance when compared to a control condition with no noise, as measured by the Karolinska Sleepiness Scale (KSS) and psychomotor vigilance task (PVT).
3. The investigators hypothesize that exposure to a blue-enriched light and a nap of up to one hour will improve subjective alertness and performance when compared to a placebo light and no nap, as measured by the Karolinska Sleepiness Scale (KSS) and psychomotor vigilance task (PVT).
4. The investigators hypothesize that sleep induced by pink noise in combination with exposure to a blue-enriched light and a nap of up to one hour will improve subjective alertness and performance when compared to a control sleep condition with no noise and a placebo light and no nap, as measured by the Karolinska Sleepiness Scale (KSS) and psychomotor vigilance task (PVT).

   PRIMARY OUTCOME MEASURES
   * Subjective alertness as measured by the 9-point Likert-type Karolinska Sleepiness Scale (KSS).
   * Objective cognitive performance as measured by the psychomotor vigilance task (PVT), a simple reaction time task with outcome measures including number of lapses (reaction time >500ms) and speed (1/reaction time).
   * Sleep architecture as measured by electroencephalography (EEG) including sleep stage at awakening, total sleep time, time in each sleep stage, sleep efficiency, and sleep onset latency.

   STATISTICAL ANALYSES To determine the impact of the interventions compared to placebo, the investigators will use a linear mixed-effects model with fixed effects of condition (intervention, control), time (test bouts post-wake-up call), condition*time interaction, and a random effect of participant. PVT lapse data (counts) will be checked for overdispersion and, if detected, a negative binomial mixed-effects model with the same factors will be used to analyze the lapse data.

   GENERAL PROTOCOL OVERVIEW Participants who pass the screening criteria and at least one week of the at-home study procedures will be asked to consent for this laboratory study. Participants will be randomized to the intervention condition and order of administration upon consent.

   Participants will not be allowed to drive to or from the lab and will be provided with a car service (taxi, Uber, Lyft, etc.) or they may arrange for a friend or family member to drop them off and pick them up.

   Participants will be maintained in a time-free environment. They will not be provided with any devices that would indicte the time. They will not be informed how long sleep and wake episodes last, nor the timing of the study activities. This is to minimize cognitive bias related to knowledge of the time of day (e.g., people may be more likely to rate themselves as sleepy during the middle of the night).

   Participants will complete hourly testing throughout their time in the lab, except during times when they are sleeping. More frequent testing may occur upon awakening from sleep. This testing will consist of the tests described below.

   Participants will be provided with three meals during their time in the lab. These meals will be provided based on the participant's dietary restrictions and personal preferences.

   A study staff member will remain with the participant at all times while the participant is awake in order to make sure the participant does not accidentally fall asleep and to monitor the participant while taking tests. The participant will be allowed to play games and talk to the study staff member when not completing study procedures.

   DETAILED PROTOCOL Participants will be asked to arrive at the laboratory three hours after their habitual wake time. They will be studied in a private room and will be monitored via a video link to the lab control room. Upon arrival, they will provide a urine sample that will be used for toxicology screening. They will then be oriented to study procedures and will complete practice tests. They will next be fitted with the EEG cap and will be provided with the sleep headphones, which will be set to deliver pink noise or silence. The room will be darkened and participant will be asked to get into bed at approximately seven hours from his/her habitual wake time and will be asked to try to sleep for four hours.

   At the end of this four-hour sleep opportunity, the participant will be awoken (if asleep) and will begin a ten-hour semi-constant posture protocol in dim light < 5 lux to collect the dim light melatonin onset (DLMO). During this time, participants will provide saliva samples every hour for the assessment of melatonin, which is a marker of the circadian rhythm. Participants will be asked to remain seated for 20 minutes prior to each sample collection because posture changes can affect the amount of melatonin measured in a sample. Testing will be scheduled for the majority of the 20 minutes prior to the sample to minimize the burden to the participant.

   Following the DLMO collection, the participant will be given a one-hour opportunity to nap or, in the placebo condition, will be asked to remain seated and engage in quiet activities under ~150 lux of light. After the rest break, the lights will either be turned on to the blue-enriched light or remain ~150 lux light depending on the randomization condition.

   After spending 25 hours in the lab, the participant's electrodes will be removed and the participant will be sent home. The participant will be advised that they can and should nap upon their return home. They will also be reminded not to drive or engage in any risky activities until they have had the opportunity to recover from the study-induced sleep deprivation.

   TESTS

   The following tests will be performed by all participants:

   Psychomotor Vigilance Task. Our benchmark performance measure will be the psychomotor vigilance test (PVT). This test has been demonstrated to be sensitive to circadian variation and sleep loss. The PVT involves a 5- or 10-minute reaction time (RT) performance test in which the participant is required to maintain the fastest possible RTs to a simple visual stimulus. The inter-stimulus interval involves a high signal rate randomly varying between 2 and 10 seconds. A variety of performance metrics showing stable circadian variation are obtained from each PVT trial including the number of lapses, optimum response times, false alarms, and the characteristics of vigilance decrement functions (i.e., slope, y-intercept) as a result of time on task. Different transforms applied to variables reduce inter-subject variability and provide stable estimates of circadian variation. PVT performance parameters have been shown to vary in synchrony with circadian phase.

   Karolinska Sleepiness Scale. The Karolinska Sleepiness Scale (KSS) is a highly sensitive subjective measurement for sleepiness. The scale consists of a nine-point Likert scale (items include: 1 = extremely alert, 2= very alert, 3 = alert, 4= rather alert, 5 = neither alert nor sleepy, 6= some signs of sleepiness, 7 = sleepy - but no difficulty remaining awake, 8= sleepy - some effort to keep awake, and 9 = extremely sleepy - fighting sleep). The KSS will be administered before a participant goes to bed, prior to the participant returning to sleep during night wakings, and in the morning upon waking.

   Visual analog scales (VAS) of mood. A series of 100-point bi-anchored mood scales including the following pairs: alert-sleepy, cheerful-miserable, calm-tense, depressed-elated, stressed-relaxed, peaceful-hostile, greedy-generous, aggressive-easygoing, lethargic-energetic. Participants are required to mark on the horizontal line to indicate how they are currently feeling.

   The Cognition Battery. Cognition is a neurocognitive assessment tool that covers the main cognitive domains (i.e., executive, episodic memory, complex cognition, social cognition, and sensorimotor speed) via 10 brief tests. The test battery was developed for the National Aeronautics and Space Administration (NASA) and specifically designed to assess cognitive functions in astronauts.

   Morphed Faces Task. Participants see a series of pictures that were created by separately morphing a neutral face with 3 different emotional faces (Angry, Happy and Sad), creating 3 different sets of pictures, each ranging from neutral to angry, happy or sad. Participants will view faces and be asked to identify each face's emotional category, as well as rate their interpretation of its intensity and valence (negative to positive).

   Self-Reported Performance Rating. Participants will be asked to rate how well they thought they performed after each test bout on a 7-point scale ranging from "extremely good" to "extremely poor."

   Karolinska Drowsiness Test (KDT). Participants will be asked to fixate on a point for three minutes, without moving or blinking (Putilov and Donskaya, 2013). The KDT provides EEG data with relatively few artifacts linked to movements or eye blinks.

   MEASURES Temperature Readings. Tympanic temperature will be monitored using a hospital-grade ear thermometer. At half-hourly intervals, trained research staff will take two temperature readings that will be recorded and plotted by study staff. If the temperature readings differ by more than one degree, a third measurement will be taken. If temperature readings reach 100 degrees Fahrenheit, the medical monitor will be consulted for further instruction. The purpose of body temperature monitoring is for us to obtain an estimate of an individual's circadian phase during the study.

   Saliva Samples. Saliva samples will be collected hourly during the DLMO portion of the study. The participant will be asked to spit into a small test tube and fill it halfway. These samples will be used to measure melatonin.

   Vital signs. Blood pressure and vital signs will be monitored every six hours, from the time the participant arrives in the lab, by a small, portable blood pressure monitor and cuff. If the participant has vital signs that fall out of the normal range, the study investigators will immediately inform the medical monitor on call. If advised by the medical monitor, the study will be ended and the investigator team will arrange for the participant to receive medical evaluation.

   STUDY POPULATION Study Population. The study population does not include astronauts. The investigators will recruit healthy participants between the ages of 18 and 60 years old.

   Sample Size. Our proposed study involves the investigation of multiple outcomes. The most well-defined and sensitive marker of sleep loss that is currently being used in spaceflight and laboratory studies is the PVT. As such, the investigators have based our power calculations on anticipated changes in PVT performance that have been associated with chronic partial sleep loss. Based on a paper describing effect sizes for changes in the PVT under different conditions of sleep loss, the investigators expect that the effect size for the change in PVT (1/RT) between conditions will be approximately 1.21 (Basner and Dinges, 2011). Using these assumptions, the investigators require 8 participants per condition (24 total) to detect a change in performance with 80% power at an alpha level of 0.05. As such, the investigators plan to recruit a minimum of 30 participants up to a maximum of 40 participants in order to account for individuals who drop out of the study or who are noncompliant with the protocol.

   INCLUSION/EXCLUSION CRITERIA

   Screening criteria for the inclusion/exclusion criteria are described in detail in the companion protocol. Participants must complete and pass all screening procedures in the screening and at-home study protocol to be eligible for this study:

   The investigators anticipate that they will study equal numbers of women and men, aged 18-65. Individuals who are pre-menopausal must be at least six months post-partum, not breastfeeding, and not planning a pregnancy in the immediate future. Individuals who are pregnant will be excluded from this study because circadian desynchrony in the form of shiftwork is associated with adverse pregnancy outcomes. Individuals who are pre-menopausal will also be offered a urinary pregnancy test during the screening process. Individuals who are on birth control medication will be able to continue their usual treatment.

   Individuals with a history of serious chronic conditions or mental illness will be excluded from the study. It is not possible to list all chronic conditions that may be exclusionary due to the number of medical conditions that would cause an individual to be ineligible. In brief, history of heart failure/disease, cancer, diabetes, seizures, respiratory diseases, sleep disorders, and Lupus are examples of conditions that would be considered exclusionary. In addition, individuals who score outside pre-defined thresholds on health screening questionnaires will also be excluded (as described previously).

   Sleep/wake history. During completion of the preliminary phone and post-consent screening questionnaires, participants will be asked a number of questions about their present, past, and future habitual sleep/wake schedule, including their habitual and prefered bed- and wake-times. Volunteers with a history of night work in the preceding 1-month period or transmeridian travel (across >2 time zones) in the three months prior to the study will be excluded. In order to exclude potential subjects with delayed or advanced sleep/wake schedule disorders from participation in the study, only subjects with a reported habitual bed time before 3 am and wake time after 4 am will be eligible for participation in the study. All volunteers will be informed that in order to be eligible for participation in the laboratory study, they will be required to maintain a regular (± 30 mins) 8.5-hour sleep schedule for up to three weeks. Individuals who are unable or unwilling to make this commitment (e.g., those with erratic schedules) will be excluded from volunteering for the study. Compliance will be monitored using a sleep/wake log and wrist activity monitor.

   Education and Language. The investigators do not anticipate studying individuals who do not understand English, given the requirement for subjects to fully understand the detailed procedures involved in the study. It is essential that all subjects be able to communicate frequently and adequately with study staff throughout the entire study.

   Pregnant People. Due to the disruption of sleep, individuals who are pregnant will be excluded from this study as a safety precaution as disrupted sleep is a potential risk factor for adverse pregnancy outcomes such as preeclampsia and preterm birth.

   Toxicology Screen. Participants will be required to provide a urine sample and complete a breathalyzer upon arrival at their first lab visit. This screen will be used to confirm that participants are free from drugs of abuse, including amphetamines, barbiturates, benzodiazepines, cocaine, marijuana, MDMA (ecstasy), methadone, methamphetamines, opiates, oxycodones, caffeine, and nicotine. The presences of any drugs of abuse will result in termination from participation in the study. Urine samples will be provided to an outside vendor for assay with a code number (no identifiable information will be included with the sample). The investigators do not expect to receive the results of this screen until after the participant has completed the first laboratory visit due to lab availability. Participants will be compensated in a pro-rated manner for any portion of the study that they completed prior to a positive toxicology screen. The coded toxicology results will be stored with the participant's other study data. The participant will be informed of the reason for study termination and will be asked to speak with the medical monitor for further guidance on their personal health status. Once a participant is excluded, the name-code link and toxicology results will be destroyed. For IRB reporting purposes, a log will be kept to describe why and how many participants were excluded from the study.

   Participants will not be excluded based on ethnicity or gender.

   STUDY EQUIPMENT All devices are commercial, off-the-shelf products with no modifications and used for the purposes of the device.

   Pink noise. Pink noise will be delivered at a volume of < 50 dB using noise canceling headphones.

   Blue-enriched lighting. Blue-enriched lighting will be delivered via a light tuned achieve 250 melanopic EDI at the angle of gaze. This level of lighting is the minimal daytime illuminance recommended for circadian health and well-being and is the required daytime illuminance level for space vehicles in NASA Standard 3001.

   iPod. Participants will be issued with an iPod Touch which includes a sleep diary, the PVT, and the KSS.

   Actigraphy. A small wristwatch-like device (Actiwatch, Philips Respironics, Murrysville, PA, USA) will be worn continuously (i.e., day and night) for one week leading up to the experimental night. The actigraph measures movement and estimates sleep and wake based on this movement.

   BrainVision EEG System. The investigators will record brain wave activity (EEG), horizontal and vertical (EOG), and muscle activity (EMG) using an electrode cap aligned to specific locations on the participant's head and face. The recordings will be monitored on a display in the Fatigue Countermeasures Laboratory Control Room. The digitized data will be downloaded onto a NASA computer and used to evaluate sleep outcomes.

   STIMULI There are two interventions that participants will experience during the study, sleep promoting (pink noise) and wake promoting (blue enriched lighting plus a nap). These will be delivered separately and together depending on randomization.

   Participants will be provided with comfortable headphones to wear throughout their daytime sleep opportunity. The headphones will deliver a continuous pink noise sound no greater than 50 decibels. Participants will be allowed to turn down the sound of the pink noise if they find it too loud. Participants will wear the headphones with no noise during the placebo condition.

   Participants randomized to the blue-enriched light and nap condition will have the blue-enriched light turned on during their nighttime stay in the lab. The light will be turned off for up to one hour during the nap. During the placebo condition, participants will have an overhead room light of ~150 lux illuminated throughout their nighttime stay in the lab. This light level reflects an older NASA standard which was used in the design of some Artemis vehicles. During the placebo condition, participants will be asked to engage in quiet activities such as reading for one hour.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals between the ages of 18 and 60

Individuals who are pre-menopausal must be at least six months post-partum, not breastfeeding, and not planning a pregnancy in the immediate future.

Exclusion Criteria:

BMI > 30

A sleep disorder of any kind

A chronic condition that could influence sleep (e.g., mood disorders, eye disorders)

A chronic condition that would interfere with data collection and/or potentially make sleep deprivation unsafe (e.g., cardiovascular disorders, diabetes, cancer)

Sensitive skin that would make electrode application intolerable

Use of medication that interferes with sleep (e.g., anti-anxiety, antihistamines, antidepressants, beta blockers)

Travel out of the time zone or stayed up all night in the past month

Individuals who are pregnant.

Individuals with a history of serious chronic conditions or mental illness. It is not possible to list all chronic conditions that may be exclusionary due to the number of medical conditions that would cause an individual to be ineligible. In brief, history of heart failure/disease, cancer, diabetes, seizures, respiratory diseases, sleep disorders, and Lupus are examples of conditions that would be considered exclusionary.

Individuals who test positive for caffeine, alcohol, nicotine, amphetamines, barbiturates, benzodiazepines, cocaine, marijuana, MDMA (ecstasy), methadone, methamphetamines, opiates, oxycodones.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Karolinska Sleepiness Scale (KSS) | Up to 120 minues
  Subjective alertness as measured by the 9-point Likert-type Karolinska Sleepiness Scale (KSS).
Psychomotor Vigilance Task (PVT) | up to 560 minutes
  Objective cognitive performance as measured by the psychomotor vigilance task (PVT), a simple reaction time task with outcome measures including number of lapses (reaction time >500ms) and speed (1/reaction time).
Electroencephalography (EEG) | up to 48 hours
  Sleep architecture as measured by electroencephalography (EEG) including sleep stage at awakening, total sleep time, time in each sleep stage, sleep efficiency, and sleep onset latency.

CONTACTS AND LOCATIONS:
Locations (1):
- NASA Ames Research Center, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barger LK, Flynn-Evans EE, Kubey A, Walsh L, Ronda JM, Wang W, Wright KP Jr, Czeisler CA. Prevalence of sleep deficiency and use of hypnotic drugs in astronauts before, during, and after spaceflight: an observational study. Lancet Neurol. 2014 Sep;13(9):904-12. doi: 10.1016/S1474-4422(14)70122-X. Epub 2014 Aug 7. PMID 25127232
- [Background] Basner M, Dinges DF. Maximizing sensitivity of the psychomotor vigilance test (PVT) to sleep loss. Sleep. 2011 May 1;34(5):581-91. doi: 10.1093/sleep/34.5.581. PMID 21532951
- [Background] Basner M, Savitt A, Moore TM, Port AM, McGuire S, Ecker AJ, Nasrini J, Mollicone DJ, Mott CM, McCann T, Dinges DF, Gur RC. Development and Validation of the Cognition Test Battery for Spaceflight. Aerosp Med Hum Perform. 2015 Nov;86(11):942-52. doi: 10.3357/AMHP.4343.2015. PMID 26564759
- [Background] Borbely AA. A two process model of sleep regulation. Hum Neurobiol. 1982;1(3):195-204. No abstract available. PMID 7185792
- [Background] Brainard GC, C. W., Ayers M, Kemp J, Warfield B, Maida J, Bowen C, Bernecker C, Lockley SW, Hanifin JP. (2013). Solid-state lighting for the International Space Station: tests of visual performance and melatonin regulation. Acta Astronautica, 92(1):21-8. https://doi.org/ http://dx.doi.org/10.1016/j.actaastro.2012.04.019
- [Background] Brown TM, Brainard GC, Cajochen C, Czeisler CA, Hanifin JP, Lockley SW, Lucas RJ, Munch M, O'Hagan JB, Peirson SN, Price LLA, Roenneberg T, Schlangen LJM, Skene DJ, Spitschan M, Vetter C, Zee PC, Wright KP Jr. Recommendations for daytime, evening, and nighttime indoor light exposure to best support physiology, sleep, and wakefulness in healthy adults. PLoS Biol. 2022 Mar 17;20(3):e3001571. doi: 10.1371/journal.pbio.3001571. eCollection 2022 Mar. PMID 35298459
- [Background] Cahill L, Gorski L, Le K. Enhanced human memory consolidation with post-learning stress: interaction with the degree of arousal at encoding. Learn Mem. 2003 Jul-Aug;10(4):270-4. doi: 10.1101/lm.62403. PMID 12888545
- [Background] Capezuti E, Pain K, Alamag E, Chen X, Philibert V, Krieger AC. Systematic review: auditory stimulation and sleep. J Clin Sleep Med. 2022 Jun 1;18(6):1697-1709. doi: 10.5664/jcsm.9860. PMID 34964434
- [Background] Caruso CC. Negative impacts of shiftwork and long work hours. Rehabil Nurs. 2014 Jan-Feb;39(1):16-25. doi: 10.1002/rnj.107. Epub 2013 Jun 18. PMID 23780784
- [Background] Czeisler CA, Duffy JF, Shanahan TL, Brown EN, Mitchell JF, Rimmer DW, Ronda JM, Silva EJ, Allan JS, Emens JS, Dijk DJ, Kronauer RE. Stability, precision, and near-24-hour period of the human circadian pacemaker. Science. 1999 Jun 25;284(5423):2177-81. doi: 10.1126/science.284.5423.2177. PMID 10381883
- [Background] Czeisler CA, Gooley JJ. Sleep and circadian rhythms in humans. Cold Spring Harb Symp Quant Biol. 2007;72:579-97. doi: 10.1101/sqb.2007.72.064. PMID 18419318
- [Background] Dorrian, J., Rogers, N. L., & Dinges, D. F. (2004). Psychomotor vigilance performance: Neurocognitive assay sensitive to sleep loss. Sleep Deprivation, 39-70.
- [Background] Ficca G, Axelsson J, Mollicone DJ, Muto V, Vitiello MV. Naps, cognition and performance. Sleep Med Rev. 2010 Aug;14(4):249-58. doi: 10.1016/j.smrv.2009.09.005. Epub 2009 Dec 3. PMID 19962331
- [Background] Flynn-Evans EE, Rueger M, Liu AM, Galvan-Garza RC, Natapoff A, Oman CM, Lockley SW. Effectiveness of caffeine and blue-enriched light on cognitive performance and electroencephalography correlates of alertness in a spaceflight robotics simulation. NPJ Microgravity. 2023 Dec 19;9(1):93. doi: 10.1038/s41526-023-00332-w. PMID 38114500
- [Background] Fucci RL, Gardner J, Hanifin JP, Jasser S, Byrne B, Gerner E, Rollag M, Brainard GC. Toward optimizing lighting as a countermeasure to sleep and circadian disruption in space flight. Acta Astronaut. 2005 May-Jun;56(9-12):1017-24. doi: 10.1016/j.actaastro.2005.01.029. PMID 15838948
- [Background] Hilditch CJ, Wong LR, Bathurst NG, Feick NH, Pradhan S, Santamaria A, Shattuck NL, Flynn-Evans EE. Rise and shine: The use of polychromatic short-wavelength-enriched light to mitigate sleep inertia at night following awakening from slow-wave sleep. J Sleep Res. 2022 Oct;31(5):e13558. doi: 10.1111/jsr.13558. Epub 2022 Jan 31. PMID 35102669
- [Background] Jones CW, Basner M, Mollicone DJ, Mott CM, Dinges DF. Sleep deficiency in spaceflight is associated with degraded neurobehavioral functions and elevated stress in astronauts on six-month missions aboard the International Space Station. Sleep. 2022 Mar 14;45(3):zsac006. doi: 10.1093/sleep/zsac006. PMID 35023565
- [Background] Kane RL, Roebuck-Spencer T, Short P, Kabat M, Wilken J. Identifying and monitoring cognitive deficits in clinical populations using Automated Neuropsychological Assessment Metrics (ANAM) tests. Arch Clin Neuropsychol. 2007 Feb;22 Suppl 1:S115-26. doi: 10.1016/j.acn.2006.10.006. Epub 2006 Nov 13. PMID 17101258
- [Background] Liu AM, Galvan-Garza RC, Flynn-Evans EE, Rueger M, Natapoff A, Lockley SW, Oman CM. Effects of caffeine and blue-enriched light on spare visual attention during simulated space teleoperation. NPJ Microgravity. 2023 Dec 19;9(1):94. doi: 10.1038/s41526-023-00299-8. PMID 38114503
- [Background] Miley AA, Kecklund G, Akerstedt T. Comparing two versions of the Karolinska Sleepiness Scale (KSS). Sleep Biol Rhythms. 2016;14(3):257-260. doi: 10.1007/s41105-016-0048-8. Epub 2016 Feb 1. PMID 28781579
- [Background] NASA Space Flight Human System Standard-Volume I: Crew Health, NASA-STD-3001, vol. 1, (2007).
- [Background] Putilov AA, Donskaya OG. Construction and validation of the EEG analogues of the Karolinska sleepiness scale based on the Karolinska drowsiness test. Clin Neurophysiol. 2013 Jul;124(7):1346-52. doi: 10.1016/j.clinph.2013.01.018. Epub 2013 Mar 6. PMID 23474052
- [Background] Okun ML, Roberts JM, Marsland AL, Hall M. How disturbed sleep may be a risk factor for adverse pregnancy outcomes. Obstet Gynecol Surv. 2009 Apr;64(4):273-80. doi: 10.1097/OGX.0b013e318195160e. PMID 19296861
- [Background] Rahman SA, Flynn-Evans EE, Aeschbach D, Brainard GC, Czeisler CA, Lockley SW. Diurnal spectral sensitivity of the acute alerting effects of light. Sleep. 2014 Feb 1;37(2):271-81. doi: 10.5665/sleep.3396. PMID 24501435
- [Background] van der Helm E, Gujar N, Walker MP. Sleep deprivation impairs the accurate recognition of human emotions. Sleep. 2010 Mar;33(3):335-42. doi: 10.1093/sleep/33.3.335. PMID 20337191
- [Background] van Rooijen R, Ploeger A, Kret ME. The dot-probe task to measure emotional attention: A suitable measure in comparative studies? Psychon Bull Rev. 2017 Dec;24(6):1686-1717. doi: 10.3758/s13423-016-1224-1. PMID 28092078
- [Background] Zhou X, Sargent C, Kosmadopoulos A, Darwent D, Dawson D, Roach GD. Do split sleep/wake schedules reduce or increase sleepiness for continuous operations? Accid Anal Prev. 2017 Feb;99(Pt B):434-439. doi: 10.1016/j.aap.2015.10.027. Epub 2015 Nov 6. PMID 26549869

DOCUMENTS (1):
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT06531733/ICF_000.pdf